CLINICAL TRIAL: NCT01892605
Title: The Clinical Application and Mechanism of Music Therapy (Mozart's Effect) on Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMU-IRB-970391
Record Dates: First submitted 2013-06-19; First posted 2013-07-04 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Seizure
Keywords: Mozart K.448; first unprovoked seizure; epileptiform discharges; music therapy; children
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- music listening, no music (Experimental): The clinical application and mechanism of music therapy The clinical application and mechanism of music therapy (Mozart's effect) on epilepsy (Mozart's effect) on epilepsy
  Interventions: Behavioral: music listening

INTERVENTIONS:
Behavioral: music listening — The treatment group listened to Mozart K.448 for eight minutes once daily before bedtime for at least six months.

SUMMARY:
Music has a long history in healing physical and mental illness. The Mozart effect was initially reported by Rauscher, Shaw, and Ky in the journal of "Nature" in the year of 1993. They examined performance on Stanford-Binet spatial tasks immediately following either 10 minutes of listening to Mozart's sonata K.448, silence, or instruction to relax. They found the performance scores were 9 point higher in Mozart-listening group than other two groups. Later, the beneficial influence of Mozart music on parkinson's disease, epilepsy, senile dementia, and attention-deficit/hyperactivity disorder was reported. However, the real neurophysiological mechanism of the influence remains unclear.

Epilepsy is a common disorder in the field of pediatric neurology. Although we had greatly advanced in develop of new anticonvulsant, thirty percent of patients with epilepsy have drug-resistance, which is associated with an increased risk of debilitating psychosocial consequences. In addition, the adverse effects of anticonvulsants are not uncommon. Few reports demonstrated that patients exposed to Mozart's music can significantly decrease in seizure frequencies and interictal epileptiform discharge. However, the case number of these studies was limited and the mechanisms of music therapy on epilepsy were not well known. In our recent studies, Mozart's music indeed decreased the epileptifrom discharge in the patients with epilepsy, particularly in the patients with generalized discharge and central discharge. On the basis of these encouraging results, we will try to investigate the neural mechanisms and clinical applications of music therapy in the following three years.

In the first year of our study, we use animal model to examine the possible mechanism of Mozart's effect. The aim of the second year study is investigation the effect of music on the cortical functions in the epileptic rat model. According to our previous study, Mozart's sonata K.448 was effective in reducing epileptiform discharge. On the basis of previous two-year results, the patients with epilepsy will be enrolled in the third year project to perform an individualized music therapy. In this study, we can provide an alternative therapy in the patients of epilepsy and investigate the possible biological mechanism of music effect.

DETAILED DESCRIPTION:
Children with first unprovoked seizure were investigated.Patients were randomly classified into treatment and control groups. They did not receive AED after their first unprovoked seizure. The treatment group listened to Mozart K.448 for eight minutes once daily before bedtime for at least six months.All of the patients received follow-up telephone calls monthly. Patients who experienced seizure recurrence were advised to begin AED treatment.

ELIGIBILITY:
Inclusion Criteria:

* children who had epileptiform discharges with first unprovoked seizure

Exclusion Criteria:

* epileptic children without epileptiform discharges

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2009-04; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
estimate seizure recurrence rate by Kaplan-Meier estimates | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Chang Lin, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Lin LC, Lee WT, Wu HC, Tsai CL, Wei RC, Mok HK, Weng CF, Lee MW, Yang RC. The long-term effect of listening to Mozart K.448 decreases epileptiform discharges in children with epilepsy. Epilepsy Behav. 2011 Aug;21(4):420-4. doi: 10.1016/j.yebeh.2011.05.015. PMID 21689988
- [Derived] Lin LC, Lee MW, Wei RC, Mok HK, Yang RC. Mozart K.448 listening decreased seizure recurrence and epileptiform discharges in children with first unprovoked seizures: a randomized controlled study. BMC Complement Altern Med. 2014 Jan 13;14:17. doi: 10.1186/1472-6882-14-17. PMID 24410973